CLINICAL TRIAL: NCT04731714
Title: Peripheral Induction of Inhibitory Brain Circuits to Treat Tourette's: Pilot
Brief Title: Median Nerve Stimulation Pilot
Acronym: MNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kevin J. Black, M.D., Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 202011092; UL1TR002345 (NIH)
Record Dates: First submitted 2021-01-13; First posted 2021-02-01 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Tourette Syndrome; Tic Disorders; Tic Disorder, Chronic Motor or Vocal
Keywords: Tourette; Tic; Transcutaneous Electric Nerve Stimulation; Median Nerve
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Tics

STUDY DESIGN:
Intervention Model Description: After screening and characterizing symptoms and other demographic and clinical features, all participants will complete two stimulation sessions, at least a week apart. These are identical except that one session uses rhythmic and one uses arrhythmic MNS with the same number of total pulses per minute. Session order is randomized and participants are blinded to order. Biological carryover effects are very unlikely. Tics before, during and after stimulation epochs are video recorded for later analysis blind to time, stimulation (on vs. off), and stimulation type (rhythmic vs. arrhythmic).
  NOTE: This study is not intended to evaluate a specific device for future use. Rather it is a study to determine the action of pulsed electrical stimulation on tic symptoms and to gain early evidence of effectiveness. This is a non-significant risk device study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The stimulation pulses will be triggered by a computer program which will provide either rhythmic or arrhythmic MNS at the same mean rate throughout a given study session. A programmer who does not interact with the participants uses a stimulation order table created by a true random number generator to select the "day 1" and "day 2" program for each participant in advance. Participants and the investigator are blind to stimulation order and stimulation type. Audiovisual recordings of tics will be rated by a reviewer who will additionally be blind to time (first vs. second stimulation session).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: rhythmic MNS, then arrhythmic MNS (Other): Participants will complete two stimulation sessions, at least a week apart. The first session involves rhythmic MNS and the second uses arrhythmic MNS.
  Interventions: Device: Rhythmic median nerve stimulation; Device: Arrhythmic median nerve stimulation
- Experimental: arrhythmic MNS, then rhythmic MNS (Other): Participants will complete two stimulation sessions, at least a week apart. The first session involves arrhythmic MNS and the second uses rhythmic MNS.
  Interventions: Device: Rhythmic median nerve stimulation; Device: Arrhythmic median nerve stimulation

INTERVENTIONS:
Device: Rhythmic median nerve stimulation — Square-wave 200 µs pulses triggered by computer at 12 Hz, at the threshold for thumb movement (expected ~2-15mA), applied to surface electrodes over the median nerve at the right wrist (conductive gel, 30 mm apart center-to-center, anode distal). This is a non-significant risk device study.
  Other Names: Rhythmic MNS
Device: Arrhythmic median nerve stimulation — Square-wave 200 µs pulses triggered by computer at random intervals with a mean rate of 12 Hz (as described in Morera Maiquez et al., 2020), at the threshold for thumb movement (expected ~2-15mA), applied to surface electrodes over the median nerve at the right wrist (conductive gel, 30 mm apart center-to-center, anode distal). This is a non-significant risk device study.
  Other Names: Arrhythmic MNS

SUMMARY:
Results from the University of Nottingham suggested that rhythmic median nerve stimulation (MNS) improves tic symptoms in Tourette syndrome (TS). The investigators will (1) provide a first replication of their study, (2) test the hypothesized electrophysiological mechanism and rule out a placebo effect as cause for the symptomatic benefit, and (3) gather information on the duration of effect after the end of stimulation and on individual characteristics that predict improvement with simulation. Completion of these Aims will give a clear go/no-go signal for a future clinical trial of chronic MNS delivered by a yet-to-be-developed wristwatch-style device.

NOTE: This study is not intended to evaluate a specific device for future use. Rather it is a study to determine the action of pulsed electrical stimulation on tic symptoms and to gain early evidence of effectiveness. This is a non-significant risk device study.

DETAILED DESCRIPTION:
Chronic tic disorders (CTD), including Tourette syndrome (TS), are associated with a substantially reduced quality of life. Medication treatments are no more than 50-60% effective in randomized controlled trials, and are often discontinued due to unacceptable side effects. Behavioral therapies require ability to participate in therapy and a specially trained therapist, but weekly visits to psychologists are impractical for many Americans, especially in rural areas. Patients strongly desire new treatment options.

In June, 2020, Stephen Jackson's group at the University of Nottingham published a fascinating report in Current Biology on a potential novel treatment for tics. The radical new idea arose from observations associating movement inhibition with 8-14 Hz activity in motor cortex. They first showed that rhythmic 12 Hz peripheral stimulation of the median nerve evoked synchronous contralateral EEG activity over primary sensorimotor cortex, whereas arrhythmic stimulation at the same mean rate did not. As hypothesized, median nerve stimulation (MNS) at 12 Hz created small but statistically significant effects on initiation of voluntary movements. Importantly, they also demonstrated that this stimulation did not meaningfully impair concentration, suggesting that the effect did not operate through simple distraction. They went on to test 10 Hz MNS in 19 TS patients, and demonstrated using blinded video ratings a significant reduction in tic number and severity during 1-minute stimulation epochs vs 1-minute no-stimulation epochs. They noted that in some participants, benefit lasted beyond the end of the stimulation epoch. Videos accompanying the publication showed dramatic benefit during MNS in some subjects. Although the authors appropriately noted the steps needed to generalize these results to clinical practice, news reports already have led a number of TS patients to contact them asking for treatment. The Nottingham group has referred such inquiries from the U.S. to me as leader of our Wash.U. Tourette Association of America (TAA) Center of Excellence.

The hypotheses of this project are that the tic benefits reported by the Nottingham investigators are replicable, that they are specific to rhythmic stimulation, which alone entrained cortical activity, rather than to a placebo effect, and that they endure past the end of stimulation.

This project (a) will replicate the Nottingham findings using identical methods, and (b) will test rhythmic MNS against a placebo treatment (arrhythmic MNS at the same mean frequency). It also will gather additional preliminary data needed for a future R01 application, including response and tolerability with longer (5-minute) stimulation blocks, and the duration of benefit after the end of a stimulation block.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-64 inclusive at initial screening visit
* Informed consent by adult subject; assent by child and informed consent by guardian
* Current Tourette's Disorder or Persistent (Chronic) Tic Disorder according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition: DSM-5
* At least 1 tic per minute (average) during the first 5-min. baseline video session on the first visit (as scored during the session by the investigator)

Exclusion Criteria:

* Unable to complete study procedures for any reason
* Has an implanted device that could be affected by electrical current
* Pregnancy known to participant or (for children) to the parent
* Known or suspected primary genetic syndrome (e.g. Down syndrome, Fragile X)
* Intellectual disability (known, or likely from history and examination)
* Head trauma with loss of consciousness for more than 5 minutes
* Significant neurologic disease, not counting TS (exceptions include febrile seizures or uncomplicated migraine)
* Severe or unstable systemic illness
* Factors (such as exaggerated signs) that in the judgment of the principal investigator make the video recording or YGTSS an inaccurate assessment of tic severity
* Judged by investigator to be unlikely to complete study procedures or to return for later visits
* Change in somatic or psychotherapeutic treatment in the 2 weeks preceding the first stimulation visit
* Planned change in somatic or psychotherapeutic treatment between the 2 stimulation visits

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Black, MD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, Movement Disorders Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Video recordings will not be shared, as they cannot feasibly be de-identified. All other individual participant data (excluding PHI) will be collected and stored on REDCap (redcap.wustl.edu) and will be shared on the Open Science Framework (OSF, at https://osf.io/mtbzf/).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol is available now (https://osf.io/mtbzf/). Statistical Analysis Plan (SAP) will be available before enrolling the first participant.
Access Criteria: Individual participant data (IPD) will be freely available under a CC0 license (Creative Commons public domain dedication, https://creativecommons.org/publicdomain/zero/1.0/).
URL: https://osf.io/mtbzf/

REFERENCES:
- [Background] Morera Maiquez B, Sigurdsson HP, Dyke K, Clarke E, McGrath P, Pasche M, Rajendran A, Jackson GM, Jackson SR. Entraining Movement-Related Brain Oscillations to Suppress Tics in Tourette Syndrome. Curr Biol. 2020 Jun 22;30(12):2334-2342.e3. doi: 10.1016/j.cub.2020.04.044. Epub 2020 Jun 4. PMID 32502412
- [Derived] Iverson AM, Arbuckle AL, Ueda K, Song DY, Bihun EC, Koller JM, Wallendorf M, Black KJ. Median Nerve Stimulation for Treatment of Tics: Randomized, Controlled, Crossover Trial. J Clin Med. 2023 Mar 27;12(7):2514. doi: 10.3390/jcm12072514. PMID 37048598
- [Derived] Iverson AM, Arbuckle AL, Ueda K, Song DY, Bihun EC, Koller JM, Wallendorf M, Black KJ. Peripheral nerve induction of inhibitory brain circuits to treat Tourette syndrome: A randomized crossover trial. medRxiv [Preprint]. 2023 Feb 6:2023.02.01.23285304. doi: 10.1101/2023.02.01.23285304. PMID 36778375
- See also: Study protocol (follow link under "Protocol") — https://osf.io/mtbzf/
- Available data/document: Individual Participant Data Set: mtbzf — https://osf.io/mtbzf/ — IPD, study protocol, SAP, and ICF will all be posted at this location.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through clinical referrals, referrals from the University of Nottingham research team, advertising and word of mouth. Recruitment began in June, 2021, with the first subject enrolled in July, 2021. Study completion was in April, 2022.
Pre-assignment Details: 2 potential participants did not meet study inclusion criteria at screening and therefore were excluded prior to study arm assignment.
Period: Overall Study
Arm/Group | Experimental: Rhythmic MNS, Then Arrhythmic MNS | Experimental: Arrhythmic MNS, Then Rhythmic MNS
Started | 16 | 16
Completed Study Visit 1 | 16 | 16
Completed Study Visit 2 | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Rhythmic MNS, Then Arrhythmic MNS | Experimental: Arrhythmic MNS, Then Rhythmic MNS | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.81 (16.81) | 31.25 (16.16) | 34.03 (16.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Tic Frequency From When MNS is Turned Off
Description: The number of tics per minute is assessed by an expert rater blind to condition and time point. Mean tic frequency was compared in on vs. off 1-minute stimulation epochs on the rhythmic MNS day. This analysis replicates that of Study 3 in the Morera Maiquez et al 2020 citation, who reported tics in the last 40 seconds of the block to minimize carryover effects. A Mixed Models Analysis was used to test statistical significance; it included a factor for possible within-day carryover effect and used a logarithmic transformation for tic count. Data reported here have been back-transformed to the number of tics in the last 40 s of the stimulation blocks.
Time Frame: During the 1-minute on and 1-minute off blocks of rhythmic MNS stimulation (total 4 blocks)
Population: All participants in the study, 4 blocks for each participant (2 on, 2 off, in random order)
Measure: Least Squares Mean (95% Confidence Interval); unit: Tic frequency (number of tics in 40 s)
Groups:
- All Participants: All participants in the study, including both those assigned to "sequence: rhythmic-arrhythmic" and those assigned to "sequence: arrhythmic-rhythmic"
Arm/Group | All Participants
Number analyzed (Participants) | 32
Tic frequency (number of tics in 40 s)
  Stimulation Off | 12.1 [9.3 to 15.8]
  Stimulation On | 8.9 [6.6 to 11.8]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.0104, Mixed Models Analysis; See publication for details

2. Primary Outcome: Change in Tic Severity From When MNS is Turned Off
Description: Severity is rated on a 5-point scale for each occurrence of any tic. The scale is the Intensity item from the Yale Global Tic Severity Scale [YGTSS], which uses integer scores from 0 (no tics) to 5 (severe intensity). Mean tic severity was compared in on vs. off 1-minute stimulation epochs on the rhythmic MNS day. This analysis replicates that of Study 3 in the Morera Maiquez et al 2020 citation.
Time Frame: During the 1-minute on and 1-minute off blocks of rhythmic MNS stimulation (total 4 blocks)
Population: All participants in the study, 4 blocks for each participant (2 on, 2 off, in random order)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 32
units on a scale
  Stimulation Off | 2.5 [2.2 to 2.7]
  Stimulation On | 2.3 [2.0 to 2.6]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.079, Mixed Models Analysis; See publication for details

3. Primary Outcome: Change in Tic Frequency During Rhythmic MNS (vs. Arrhythmic MNS)
Description: The number of tics per minute is assessed by an expert rater blind to condition and time point. Change in tic frequency from baseline (stimulation off) is compared between 5-minute MNS-on epochs on the rhythmic vs. the arrhythmic day. Subjects who do not complete both stimulation visits will not be included in this analysis. The hypothesized change is greater improvement (off to on) with rhythmic vs. arrhythmic stimulation. This analysis includes the first six 5-minute blocks on each MNS day (i.e., the blocks that all participants complete). MNS was administered throughout blocks 6 and 8 only. Tic frequency in block 0 (baseline, before any stimulation) on the same day was a covariate in the statistical model.
Time Frame: During 5-minute MNS stimulation on or off blocks 0, 5, 6, 7, 8 and 9
Population: All participants in the study
Measure: Least Squares Mean (95% Confidence Interval); unit: Tic frequency (number of tics in 5 min.)
Arm/Group | All Participants
Number analyzed (Participants) | 32
Tic frequency (number of tics in 5 min.)
  Arrhythmic Block 5 | 85.8 [69.2 to 102.4]
  Arrhythmic Block 6 | 63.3 [46.5 to 80.2]
  Arrhythmic Block 7 | 74.2 [57.3 to 91.2]
  Arrhythmic Block 8 | 57.7 [40.8 to 74.5]
  Arrhythmic Block 9 | 65.0 [48.4 to 81.6]
  Rhythmic Block 5 | 85.9 [69.7 to 102.1]
  Rhythmic Block 6 | 61.8 [45.4 to 78.2]
  Rhythmic Block 7 | 67.5 [51.0 to 83.9]
  Rhythmic Block 8 | 57.6 [41.2 to 74.0]
  Rhythmic Block 9 | 68.4 [52.2 to 84.7]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.9222, Mixed Models Analysis; See publication for details

4. Primary Outcome: Change in Tic Severity During Rhythmic MNS (vs. Arrhythmic MNS)
Description: Overall tic severity for each 5-minute block is rated once on a 5-point scale by an expert blind to condition and time point. The scale is the Intensity item from the Yale Global Tic Severity Scale [YGTSS], which uses integer scores from 0 (no tics) to 5 (severe intensity). Change in tic severity from baseline (stimulation off) is compared between 5-minute MNS-on epochs on the rhythmic vs. the arrhythmic day. Subjects who do not complete both stimulation visits will not be included in this analysis. The hypothesized change was greater improvement (off to on) with rhythmic vs. arrhythmic stimulation. This analysis includes the first six 5-minute blocks on each MNS day (i.e., the blocks that all participants complete). MNS was administered throughout blocks 6 and 8 only. Tic frequency in block 0 (baseline, before any stimulation) on the same day was a covariate in the statistical model.
Time Frame: During 5-minute MNS stimulation on or off blocks 0, 5, 6, 7, 8 and 9
Population: All participants in the study
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 32
units on a scale
  Arrhythmic Block 5 | 3.4 [3.1 to 3.6]
  Arrhythmic Block 6 | 3.2 [2.9 to 3.5]
  Arrhythmic Block 7 | 3.4 [3.1 to 3.6]
  Arrhythmic Block 8 | 3.0 [2.7 to 3.3]
  Arrhythmic Block 9 | 3.1 [2.8 to 3.3]
  Rhythmic Block 5 | 3.3 [3.0 to 3.6]
  Rhythmic Block 6 | 3.2 [2.9 to 3.4]
  Rhythmic Block 7 | 3.2 [2.9 to 3.5]
  Rhythmic Block 8 | 3.1 [2.8 to 3.3]
  Rhythmic Block 9 | 3.1 [2.8 to 3.3]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.7995, Mixed Models Analysis; See publication for details

5. Secondary Outcome: Change in Tic Severity After MNS Ends
Description: We compared the change in tic frequency from baseline, during each 1-minute-long period following the end of stimulation. Here baseline means the tic frequency during the last 5 minutes of MNS from the same day (block 8). Last observation carried forward was used for participants who had less than 20 minutes of data following block 8.
Time Frame: up to 20 minutes after the end of stimulation at each study visit up to 1 month
Population: All participants in the study
Measure: Median (Inter-Quartile Range); unit: Tic frequency (tics per minute)
Arm/Group | All Participants
Number analyzed (Participants) | 32
Tic frequency (tics per minute)
  Final Block Of Stimulation, rhythmic days | 7.1 [3.95 to 12.4]
  20 minutes after stimulation, rhythmic days | 12 [5 to 17.75]
  Final Block Of Stimulation, arrhythmic days | 8 [3.7 to 18.7]
  20 minutes after stimulation, arrhythmic days | 10 [5 to 22]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.3140, Friedman Test — rhythmic days; See publication for further details
Statistical Analysis 2: Comparison: All Participants; Test type: Other; p = 0.239, Friedman Test — arrhythmic days; See publication for further details

6. Secondary Outcome: CGI-I, Participant
Description: Clinical Global Impression of Improvement (CGI-I), rated by participant. The CGI-I is a 7-point scale ranging from 1 = very much improved to 7 = very much worse.
Time Frame: 5-25 minutes after the end of stimulation at each study visit up to 1 month
Population: All participants in the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 32
units on a scale
  Rhythmic Day | 2.69 (1.03)
  Arrhythmic Day | 2.39 (0.99)

7. Secondary Outcome: CGI-I, Investigator
Description: Clinical Global Impression of Improvement (CGI-I), rated by investigator. The CGI-I is a 7-point scale ranging from 1 = very much improved to 7 = very much worse.
Time Frame: 5-25 minutes after the end of stimulation at each study visit up to 1 month
Population: All participants in the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 32
units on a scale
  Rhythmic Day | 2.41 (0.91)
  Arrhythmic Day | 2.56 (1.01)

8. Secondary Outcome: Rating of Therapeutic Effect Using the CGI Efficacy Index
Description: Participant rates peak improvement experienced during the visit using the 4-point scale of the CGI (Unchanged or worse; Minimal - Slight improvement that doesn't decrease the overall impact of symptoms*; Moderate - Decided improvement. Partial remission of symptoms; Marked - Vast improvement. Complete or nearly complete remission of all symptoms). * = "Minimal" option anchor text slightly edited from original. The number provided is the number of participants who rated each visit as moderate or marked.
Time Frame: 5-25 minutes after the end of stimulation at each study visit up to 1 month
Population: All participants in the study
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 32
Participants
  Rhythmic Day | 20
  Arrhythmic Day | 23

9. Secondary Outcome: VAS (Visual Analog Scale) Rating of Premonitory Urge Severity
Description: Participant rates the maximal severity of any premonitory urges over the preceding minute, from 0=no premonitory urge to 100=maximally uncomfortable premonitory urge, using a Visual Analog Scale.
Time Frame: At the end of each 5-min. MNS on or off block through block 9, at each study visit
Population: All participants in the study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 32
units on a scale
  Arrhythmic Block 5 | 50.1 [43.7 to 56.6]
  Arrhythmic Block 6 | 36.5 [30.0 to 43.1]
  Arrhythmic Block 7 | 43.0 [36.5 to 49.6]
  Arrhythmic Block 8 | 32.0 [25.4 to 38.7]
  Arrhythmic Block 9 | 38.4 [31.9 to 45.0]
  Rhythmic Block 5 | 50.3 [43.8 to 56.8]
  Rhythmic Block 6 | 34.1 [27.6 to 40.7]
  Rhythmic Block 7 | 45.5 [39.0 to 52.1]
  Rhythmic Block 8 | 32.8 [26.3 to 39.4]
  Rhythmic Block 9 | 40.5 [34.1 to 47.0]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.8844, Mixed Models Analysis; See publication for details

10. Secondary Outcome: Rating of Discomfort Using the CGI Efficacy Index (Edited)
Description: Participant rates peak discomfort experienced during the visit using the 4-point scale of the CGI: "Overall, today, how much DISCOMFORT did the stimulation cause? If discomfort is the wrong word, please substitute any negative effects or side effects of stimulation. (No discomfort; Discomfort noticeable, but not severe enough to concern me or to turn it off; Enough discomfort, impairment of functioning or social embarrassment that I would only keep it on if the benefit was considerable; Caused discomfort, impairment of functioning or social embarrassment to a degree that any treatment benefit was not worth leaving it on). The number provided is the number of visits where discomfort is rated as none or minimal.
Time Frame: 5-25 minutes after the end of stimulation at each study visit up to 1 month
Population: All study visits (2 per participant)
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | All Participants
Number analyzed (Participants) | 32
Number analyzed (Visits) | 64
Visits | 57

11. Secondary Outcome: Blindedness Assessment
Description: Participants guess at each study visit whether they received the active or sham MNS condition, and rate their certainty for that guess on a 0-3 scale (0 = pure guess, 3 = certain). The number reported here is the number of visits for which the participant guessed correctly (active vs. sham MNS).
Time Frame: 5-25 minutes after the end of stimulation at each study visit up to 1 month
Population: One guessed treatment assignment for each study visit (1 guess per visit, 2 visits per participant)
Measure: Count of Units; unit: treatment guess on a given study visit
Units Other Than Participants: treatment guess on a given study visit
Arm/Group | All Participants
Number analyzed (Participants) | 32
Number analyzed (treatment guess on a given study visit) | 64
treatment guess on a given study visit
  Guessed correctly | 30
  Guessed incorrectly | 34
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.73, binomial; One-sided

ADVERSE EVENTS:
Time Frame: From enrollment through final study visit, up to 1 month
Groups:
- Experimental: Rhythmic MNS: Rhythmic median nerve stimulation: Square-wave 200 µs pulses triggered by computer at 12 Hz, at the threshold for thumb movement (expected ~2-15mA), applied to surface electrodes over the median nerve at the right wrist (conductive gel, 30 mm apart center-to-center, anode distal). This is a non-significant risk device study.
- Experimental: Arrhythmic MNS: Arrhythmic median nerve stimulation: Square-wave 200 µs pulses triggered by computer at random intervals with a mean rate of 12 Hz (as described in Morera Maiquez et al., 2020), at the threshold for thumb movement (expected ~2-15mA), applied to surface electrodes over the median nerve at the right wrist (conductive gel, 30 mm apart center-to-center, anode distal). This is a non-significant risk device study.
Arm/Group | Experimental: Rhythmic MNS | Experimental: Arrhythmic MNS
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 4/32 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Rhythmic MNS (N=32) | Experimental: Arrhythmic MNS (N=32)
(Nervous system disorders) | 2 | 3 — These participants did not specify the discomfort but rated its severity as more than mild.
Headache (Nervous system disorders) | 1 | 0 — Participant description was "like an ocular migraine without the aura."
Itch (Nervous system disorders) | 1 | 0 — Participant description was "Itching / stinging under the electrode."

LIMITATIONS AND CAVEATS:
We did not test other variations on MNS, so we cannot address the specificity of the median nerve (vs. any other peripheral nerve), the specificity of 10-12 Hz as the stimulation frequency, or whether there is a lateral preference for MNS benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT04731714/Prot_SAP_000.pdf